CLINICAL TRIAL: NCT05527184
Title: A Phase 1, First-in-Human, Open-Label, Dose-Escalation and Expansion Study of IMGN151 (Anti-FRα Antibody-drug Conjugate) in Adult Patients With Recurrent Gynaecological Cancers
Brief Title: First in Human Study of IMGN151 in Recurrent Gynaecological Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMGN151-1001; 2023-506842-22 (Other: EU CT)
Record Dates: First submitted 2022-08-23; First posted 2022-09-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer; High Grade Serous Adenocarcinoma of Ovary; Primary Peritoneal Carcinoma; Fallopian Tube Cancer; Cervical Cancer
Keywords: Antibody Drug Conjugate; Platinum-Resistant; Recurrent
MeSH Terms: conditions — Endometrial Neoplasms; Fallopian Tube Neoplasms; Uterine Cervical Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMGN151 (Experimental): IMGN151 is administered via intravenous (IV) infusion on Day 1 of Cycle 1 every 3-week cycle (Q3W).
  Interventions: Drug: IMGN151

INTERVENTIONS:
Drug: IMGN151 — IMGN151 is an antibody-drug conjugate (ADC).

SUMMARY:
IIMGN151-1001 is a Phase 1, first in human, open-label dose-escalation, optimization, and expansion study designed to characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity, and preliminary antitumor activity of IMGN151 in adult participants with recurrent endometrial cancer; recurrent, high-grade serous epithelial ovarian, fallopian tube, and primary peritoneal cancers; or recurrent cervical cancers. All participants will be, in the opinion of the investigator, appropriate for nonplatinum single-agent therapy for their next line of therapy.

DETAILED DESCRIPTION:
Participants may continue on study drug based on clinical benefit until disease progression, adverse event (AE) requiring discontinuation, withdrawal of consent, physician decision, or other discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
2. Dose-Escalation Phase: Recurrent endometrial cancer or high-grade serous epithelial ovarian, fallopian tube, and primary peritoneal cancer (EOC) and who have exhausted appropriate standard-of-care therapy.
3. Dose Optimization: Platinum-resistant, high-grade serous EOC (PROC) with no previous folate receptor alpha (FRα)-directed therapy. Participants with PROC will have had no more than 5 prior lines of therapy, with no more than 2 prior therapies since development of platinum resistance.
4. Expansion Phase:

   1. For Cohort A, recurrent endometrial cancer (high-grade endometrioid or serous histology only) with 1-3 prior lines of therapy.
   2. For Cohort B, PROC with no previous FRα-directed therapy and no more than 5 prior lines of therapy, with no more than 2 prior therapies since development of platinum resistance.
   3. For Cohort C, PROC with previous FRα-directed therapy with at least one intervening anticancer therapy between prior FRα-directed therapy and IMGN151.
   4. For Cohort D, EOC of one of the following histologies: carcinosarcoma, endometrioid, and low-grade serous carcinoma and have exhausted appropriate standard-of-care therapy.
   5. For Cohort E, cervical cancer including the following histologies: squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma with 1-4 prior lines of therapy.
   6. For participants with cervical cancer with Combined Positive Score (CPS) > 1 or with endometrial cancer, prior checkpoint inhibitor therapy, alone or in combination, is required if available locally and medically appropriate.
5. Evaluable lesions

   1. Dose-Escalation Phase: Participants may have radiologically evaluable or nonevaluable disease.
   2. Dose Optimization and Expansion Phase: Participants must have at least 1 lesion that meets the definition of measurable disease by RECIST v1.1 (radiologically measured by the investigator).
6. Willing to provide an archival tumor tissue block or slides or to undergo a procedure to obtain a new biopsy using a low-risk, medically routine procedure.
7. Participants must have stabilized or recovered (Grade 1 or baseline) from all prior therapy-related toxicities (except alopecia or hemoglobin within 10 days before Cycle 1 Day 1).
8. Participants must have completed any major surgery at least 4 weeks prior to first dose of IMGN151 and have recovered or stabilized from the side effects of prior surgery prior to first dose of IMGN151.
9. Participants must have adequate organ and bone marrow function.

Exclusion Criteria:

1. Participants with ovarian cancer with histologies including clear cell, mucinous, or borderline ovarian tumor.

   1. With the exception of participants enrolled in Cohort D, participants with ovarian cancer with histologies including endometrioid, sarcomatous histology, mixed tumors containing any of the above histologies, as well as low-grade serous carcinoma.
   2. For Cohort A, participants with endometrial cancer with histologies other than high-grade serous or high-grade endometrioid.
   3. For Cohort E, participants with cervical cancer with histologies other than adenocarcinoma, squamous cell carcinoma, and adenosquamous carcinoma.
2. For Cohort B and Dose Optimization: participants with primary platinum refractory ovarian cancer, defined as disease progression on or within 3 months completion of first platinum-based treatment.
3. Radiation therapy of > 20% of the potential bone marrow
4. Participants with > Grade 1 peripheral neuropathy per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
5. Participants with the following ocular history and/or concurrent disorders:

   1. Active or chronic corneal epithelial disorders other than non-confluent superficial keratopathy/keratitis, including confluent superficial punctate keratopathy/keratitis (SPK) not expected to resolve to non-confluence or better within the screening window with standard-of-care intervention
   2. History of corneal transplantation
   3. Undergoing active postoperative management for refractive surgery, cataract surgery, corneal cross-linking, or corneal complications of surgery
   4. Active or chronic clinically significant (≥ Grade 3) corneal disorders (for example, Fuch's dystrophy or neurotrophic keratitis)
   5. Active ocular conditions requiring ongoing treatment/monitoring, such as glaucoma, which is not adequately controlled with medication or surgery, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, presence of papilledema, an ocular condition with high risk of retinal detachment
   6. Monocular vision with visual acuity in the worse-seeing eye (worse than 20/200 or visual fields less than 20 degrees)
6. Serious concurrent illness or clinically relevant active infection.
7. A history of multiple sclerosis or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome)
8. Participants with clinically significant cardiac disease.
9. A history of hemorrhagic or ischemic stroke within 6 months before enrollment
10. A history of cirrhotic liver disease (Child-Pugh Class B or C)
11. Participants with evidence of pneumonitis on baseline imaging or Participants with a previous clinical diagnosis of noninfectious interstitial lung disease (ILD), including noninfectious pneumonitis
12. Participants with prior hypersensitivity to monoclonal antibodies (mAb)
13. Females who are pregnant or breastfeeding
14. For Dose Optimization and Expansion Phase: Participants who received a prior FRα-targeting agent, with the exception of participants enrolled in the prior FRα-targeting agent, ovarian cancer cohort (Cohort C).
15. Untreated or symptomatic central nervous system metastases
16. A history of other malignancy within 3 years before enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 3 years
Number of Participants With Dose-limiting Toxicities (DLTs) | Day 21 of Cycle 1 (Cycle length = 3 weeks)
Recommended Dose of IMGN151 Monotherapy | Up to approximately 2 years

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of IMGN151 | Up to approximately 3 years
Time to Reach Cmax (Tmax) of IMGN151 | Up to approximately 3 years
Area Under the Curve From Time 0 to Infinity (AUC0-inf) of IMGN151 | Up to approximately 3 years
Number of Participants With Treatment-emergent Anti-drug Antibodies (ADAs) | Up to approximately 3 years
Objective Response Rate (ORR) | Up to approximately 3 years
  ORR is defined as the percentage of participants with best response of complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
Duration of Response (DOR) | Up to approximately 3 years
  DOR is defined as the time from initial response (CR or PR) until radiological progressive disease (PD), as assessed by the investigator, or death, whichever occurs first per RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (58):
- United States (32):
  - University of Alabama at Birmingham /ID# 269045, Birmingham, Alabama
  - City of Hope National Medical Center /ID# 269036, Duarte, California
  - Moores Cancer Center /ID# 269040, La Jolla, California
  - University of California Los Angeles Medical Center /ID# 269037, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian /ID# 269047, Newport Beach, California
  - UCHSC Anschultz Cancer Pavilion /ID# 269056, Aurora, Colorado
  - AdventHealth Celebration /ID# 269030, Kissimmee, Florida
  - Mount Sinai Medical Center /ID# 269050, Miami, Florida
  - Miami Cancer Institute at Baptist Health /ID# 269041, Miami, Florida
  - Florida Cancer Specialists- Sarasota Cattlemen /ID# 269055, Sarasota, Florida
  - University of Chicago Medical Center /ID# 269028, Chicago, Illinois
  - Massachusetts General Hospital /ID# 278119, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 269039, Boston, Massachusetts
  - Karmanos Cancer Institute - Detroit /ID# 269052, Detroit, Michigan
  - University of Mississippi Medical Cancer Center /ID# 269046, Jackson, Mississippi
  - Washington University School of Medicine - St. Louis /ID# 269048, St Louis, Missouri
  - Holy Name Medical Center /ID# 269051, Teaneck, New Jersey
  - Roswell Park Cancer Institute /ID# 269043, Buffalo, New York
  - Long Island Jewish Medical Center /ID# 269035, New Hyde Park, New York
  - Columbia University Irving Medical Center /ID# 269033, New York, New York
  - University of Rochester Medical Center /ID# 269044, Rochester, New York
  - University of North Carolina Medical Center /ID# 269027, Chapel Hill, North Carolina
  - Atrium Health Levine Cancer Institute /ID# 269049, Charlotte, North Carolina
  - The Ohio State University Comprehensive Cancer Center /ID# 269026, Columbus, Ohio
  - OU Health - Stephenson Cancer Center /ID# 269025, Oklahoma City, Oklahoma
  - University of Pennsylvania /ID# 269042, Philadelphia, Pennsylvania
  - West Penn Hospital /ID# 269054, Pittsburgh, Pennsylvania
  - Women & Infants Hospital /ID# 269032, Providence, Rhode Island
  - Sanford Cancer Center /ID# 269038, Sioux Falls, South Dakota
  - Tennessee Oncology Nashville /ID# 269029, Nashville, Tennessee
  - MD Anderson Houston /ID# 269057, Houston, Texas
  - University of Virginia /ID# 269053, Charlottesville, Virginia
- Monash Health - Monash Medical Centre /ID# 268971, Perth, Western Australia, Australia
- Belgium (2):
  - Hôpital Vivalia De Libramont /ID# 268979, Libramont-Chevigny, Luxembourg
  - Universitair Ziekenhuis Leuven /ID# 268977, Leuven, Vlaams-Brabant
- Canada (4):
  - Cross Cancer Institute /ID# 268984, Edmonton, Alberta
  - BC Cancer - Kelowna /ID# 268983, Kelowna, British Columbia
  - Centre Hospitalier De L'Universite De Montreal - Hopital Saint-Luc /ID# 268982, Montreal, Quebec
  - Centre Hospitalier Universite De Sherbrooke - Hôtel-Dieu Hospital /ID# 268981, Sherbrooke, Quebec
- France (5):
  - Institut de Cancerologie de Ouest /ID# 268997, Saint-Herblain, Pays de la Loire Region
  - Centre Antoine-Lacassagne /ID# 269000, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre Leon Berard /ID# 268993, Lyon, Rhone
  - Hospices Civils de Lyon - Centre Hospitalier Lyon-Sud /ID# 268996, Pierre-Bénite, Rhone
  - Institut Gustave Roussy /ID# 268994, Villejuif, Île-de-France Region
- DKD Helios Klinik Wiesbaden /ID# 269011, Wiesbaden, Germany
- Mater Misericordiae University Hospital /ID# 269013, Dublin, Ireland
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 269020, Rome, Roma
  - Azienda Ospedaliero Universitaria delle Marche /ID# 269018, Ancona
- Netherlands (3):
  - Erasmus Medisch Centrum /ID# 269022, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen /ID# 269023, Groningen
  - Universitair Medisch Centrum Utrecht /ID# 269024, Utrecht
- Spain (7):
  - Institut Català d'Oncologia (ICO) - Badalona /ID# 268990, Badalona, Barcelona
  - Hospital Universitario Reina Sofia /ID# 269656, Córdoba, Cordoba
  - Hospital Universitario Vall de Hebron /ID# 268986, Barcelona
  - Hospital MD Anderson Cancer Center Madrid /ID# 268991, Madrid
  - Hospital Universitario Ramón y Cajal /ID# 268992, Madrid
  - Hospital Universitario La Paz /ID# 268987, Madrid
  - Hospital Clínico Universitario de Valencia /ID# 268988, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=IMGN151-1001